CLINICAL TRIAL: NCT06208904
Title: The Involvement of the Gut Hormone GIP in the Pathophysiology of Post Prandial Hypotension
Acronym: GA-21
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, lise wilki-kurtzhals, Medical Doctor and PhD student, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GIPR-Ant-21
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: PostPrandial Hypotension
Keywords: Postprandial hypotension; Glucose-dependent insulinotropic polypeptide; GIP; GIP receptor antagonist; GIP(3-30)NH2
MeSH Terms: interventions — gastric inhibitory polypeptide (3-30)-amide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GIPRA (Glucose-dependent Insulinotropic Polypepetide Receptor Antagonist) (Experimental): Intravenous infusion of GIP(3-30)NH2 in a concentration of 1,000 pmol/kg/min
  Interventions: Other: Intravenous infusion of GIPRA
- Saline (Placebo Comparator): Intravenous infusion of isotonic saline 9 mg/ml added 0,5% human serum albumin
  Interventions: Other: Intravenous infusion of saline

INTERVENTIONS:
Other: Intravenous infusion of GIPRA — Intravenous infusion of GIP(3-30)NH2 in a concentration of 1,000 pmol/kg/min during experimental days
  Other Names: GIP(3-30)NH2
  Arms: GIPRA (Glucose-dependent Insulinotropic Polypepetide Receptor Antagonist)
Other: Intravenous infusion of saline — Intravenous infusion of isotonic saline 9 mg/ml added 0,5% human serum albumin during experimental days
  Other Names: Placebo (Saline)
  Arms: Saline

SUMMARY:
The present study investigates the involvement of the gut hormone glucose-dependent insulinotropic polypeptide (GIP) in the pathophysiology of postprandial hypotension (PPH)

DETAILED DESCRIPTION:
The study is an exploratory, randomised, placebo-controlled, double-blind crossover study comprising two experimental days with an infusion of the GIP receptor antagonist, GIP(3-30)NH2 (NH2 is the aminogroup), and placebo (saline) during a 180-minute mixed meal test (MMT). Eighteen participants, men and women, with MMT confirmed PPH will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years
2. History of PPH-related symptoms like dizziness, lightheadedness, palpitations, or fainting after meal ingestion
3. Informed consent

Exclusion Criteria:

1. Not fulfilling the PPH diagnosis during the mixed meal test or during the test meal with increased (+25%) number of calories
2. Treatment with antihypertensives
3. Treatment with SNRI (Serotonin and Noradrenalin Reuptake Inhibitor) or treatment within three months before screening visit
4. Allergy or intolerance to ingredients included in the mixed meal
5. Any ongoing medication that the investigator evaluates would interfere with trial participation
6. Any physical or psychological condition that the investigator evaluates would interfere with trial participation, including any acute or chronic illnesses
7. Anaemia (haemoglobin below normal range <7.3 mmol/L for women and <8.3 mmol/L for men)
8. Moderate to severe loss of kidney function (estimated glomerular filtration rate (eGFR) <45 ml/min/1.73 m2) at screening
9. Known liver disease (except for simple steatosis) and/or elevated plasma alanine aminotransferase (ALT) > three times the upper limit of normal at screening
10. Any concomitant disease or treatment that, at the discretion of the investigators, might jeopardize the participant's safety during the trial
11. Alcohol/drug abuse as per discretion of the investigators
12. Pregnancy or breastfeeding
13. Participation in any other clinical trial during study period
14. Mental incapacity or language barriers that preclude adequate understanding or cooperation or unwillingness to comply with trial requirements or pr discretion of the investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Nadir systolic blood pressure (SBP) (mmHg) | -45-0 minutes
  Baseline
Nadir systolic blood pressure (mmHg) | 0-180 minutes
  Nadir and time to nadir

SECONDARY OUTCOMES:
Occurrence of PPH | 0-180 minutes
  (Yes/No) PPH is defined as either a drop in SBP >20 mmHg from baseline or SBP <90 mmHg
Systolic blood pressure (mmHg) | -45-0 minutes
  Baseline
Systolic blood pressure (mmHg) | 0-180 minutes
  Peak, nadir and iAUC (incremental area under the curve)
Diastolic blood pressure (mmHg) | -45-0 minutes
  Baseline
Diastolic blood pressure (mmHg) | 0-180 minutes
  Peak, nadir and iAUC
Heart rate (beats/min) | -45-0 minutes
  Baseline
Heart rate (beats/min) | 0-180 minutes
  Peak, nadir and iAUC
Stroke volumen (ml) | -45-0 minutes
  Baseline
Stroke volumen (ml) | 0-180 minutes
  Peak, nadir and iAUC
Cardiac output (l/min) | -45-0 minutes
  Baseline
Cardiac output (l/min) | 0-180 minutes
  Peak, nadir and iAUC

OTHER OUTCOMES:
Plasma glucose | -45-0 minutes
  Baseline
Plasma glucose | 0-180 minutes
  Peak, nadir and iAUC
Gastric emptying rate | -45-0 minutes
  Plasma acetaminophen, baseline
Gastric emptying rate | 0-180 minutes
  Plasma acetaminophen, peak and time to peak
Plasma GIP(3-30)NH2 | -45-0 minutes
  Baseline
Plasma GIP(3-30)NH2 | 0-180 minutes
  Peak and iAUC

CONTACTS AND LOCATIONS:
Overall Officials: Lise Wilki-Kurtzhals, Principal Investigator — University Hospital, Gentofte, Copenhagen
Locations (1):
- Center for Clinical Metabolic Research, Copenhagen, Hellerup, Denmark